CLINICAL TRIAL: NCT06940141
Title: A Phase 2, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Rademikibart as an Add-on Treatment for Acute Exacerbation in Adult and Adolescent Participants With Asthma and Type 2 Inflammation
Brief Title: Rademikibart Add-on Treatment of an Acute Asthma Exacerbation (Seabreeze STAT Asthma)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-201-206
Record Dates: First submitted 2025-04-03; First posted 2025-04-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Asthma Acute
Keywords: Acute exacerbation; Asthma; Asthma exacerbation; CBP-201; Rademikibart; Connect Biopharma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Rademikibart (Experimental)
  Interventions: Combination Product: Rademikibart in prefilled syringe
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo in prefilled syringe

INTERVENTIONS:
Combination Product: Rademikibart in prefilled syringe — Participants receive 600 mg (4mL) of rademikibart administered subcutaneously.
  Other Names: CBP-201
  Arms: Rademikibart
Drug: Matching placebo in prefilled syringe — Participants receive 4mL of placebo matched to rademikibart administered subcutaneously.
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, multicenter study in adult and adolescent participants with asthma and type 2 inflammation

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, interventional trial in participants with an acute asthma exacerbation with type 2 inflammation to compare rademikibart plus standard therapy to standard therapy alone (plus placebo), targeting an acute asthma exacerbation in the urgent healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma with duration of ≥12 months.
* Currently receiving treatment with low, medium, to high dose ICS in combination with at least 1 additional asthma controller medication.
* Must have experienced at least 1 asthma exacerbation requiring the use of systemic corticosteroids.
* For participants in a stable condition, must have a documented historical peripheral blood eosinophil count of ≥250 cells/μL and/or FeNO ≥ 25 ppb.
* Current acute asthma exacerbation requiring an urgent healthcare visit for treatment.
* Peripheral blood eosinophil count of ≥300 cells/µL as part of the assessment of an index acute asthma exacerbation.
* Requires systemic corticosteroid as SoC in the urgent healthcare setting to treat the current acute asthma exacerbation.
* FEV1 ≥30% predicted.

Exclusion Criteria:

* Regular use of immunosuppressive medication.
* Unstable ischemic heart disease, cardiomyopathy, heart failure, uncontrolled hypertension.
* Current or former smoker, has a smoking history including: If <30 years old: Smoked for ≥5 pack-years; If ≥30 years old: Smoked for ≥10 pack-years
* COPD and other clinically significant pulmonary disease other than asthma.
* Known or suspected history of immunosuppression.
* History of known immunodeficiency disorder or hepatitis B or C.
* History of alcohol abuse and/or drug abuse.
* Recent history of cancer except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy or other malignancies treated with apparent success with curative therapy.
* Female participant who is pregnant, lactating or breast-feeding, or has a positive urinary β hCG test prior to randomization.
* Recent receipt of any marketed nonbiologic drug that modulates type 2 cytokines (eg, suplatast tosilate).
* Recent receipt of any marketed biologic drug or any investigational biologic for asthma or other diseases.
* Recent live, attenuated vaccinations or planned live, attenuated vaccinations during the trial.
* Participants that have been recently treated with bronchial thermoplasty.
* Recent treatment with OCS and/or hospitalization for an exacerbation of asthma.
* Recent receipt of any investigational nonbiologic drug.
* A recent chest X-ray or computed tomography (CT) with findings that are inconsistent for an asthmatic population.

The above inclusion and exclusion criteria are not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Treatment failure rate within 28 days after randomization | 28 days
  Treatment failure is defined as death due to any cause, (re)admission to a hospital for asthma, ED (re)visit or unscheduled medical visit for worsening of asthma symptoms, or the necessity to intensify pharmacologic treatment (including second course of systemic steroids for asthma exacerbation) within 28 days after randomization.

SECONDARY OUTCOMES:
Rate of new asthma exacerbations in the 28 days after randomization | 28 days
Time to the first new asthma exacerbation in the 28 days after randomization | 28 days
Mean change from baseline (CFB) in morning/evening asthma symptom score | Week 1, Week 2, and Week 4
Mean change from baseline (CFB) in nocturnal awakenings (e-diary) | Week 1, Week 2, and Week 4
Absolute CFB in post-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) | Day 3, Week 1, and Week 4
Incidence of adverse events (AEs), including serious adverse events (SAEs), adverse event of special interest (AESIs), and drug-induced liver injury (DILI) reported | 56 days
Incidence of unanticipated adverse device effects (UADEs) | 56 days
Incidence of injection site reactions | 56 days

CONTACTS AND LOCATIONS:
Locations (41):
- United States (14):
  - Amicis Research Center, Valencia, California
  - Synergy Healthcare, Bradenton, Florida
  - Pharmax Research of South Florida, Inc., Miami, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Health Synergy Clinical Research, LLC, West Palm Beach, Florida
  - Primeway Clinical Research Group, Fayetteville, Georgia
  - Pivotal Research Solutions, Stonecrest, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Inquest Clinical Research, Baytown, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine, Denison, Texas
  - DCT- McAllen Primary Care Research, LLC dba Discovery Clinical Trials, McAllen, Texas
- Argentina (5):
  - STAT Research, Caba, Buenos Aires
  - Centro respiratorio Infantil, Rosario, Santa Fe Province
  - INECO Neurociencias Oroño, Rosario, Santa Fe Province
  - Investigaciones en Patologias Respiratorias SRL, San Miguel de Tucumán, Tucumán Province
  - INSARES, Mendoza
- Australia (4):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St George Hospital, South Eastern Sydney Local Health District, Kogarah, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
- Georgia (6):
  - "NCTLD National Center for Tuberculosis and Lung Disease" JSC, Tbilisi
  - LLC "Israel-Georgian Medical Research Clinic Healthycore", Tbilisi
  - Acad. Chapidze Emergency Cardiology Center LLC, Tbilisi
  - Caucasus Medical Center, Tbilisi
  - LLC Diacor, Tbilisi
  - Raymann, LLC, Tbilisi
- Serbia (5):
  - Clinical Hospital Center "Dragisa Misovic - Dedinje", Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
  - Institute for Pulmonary Diseases and Tuberculosis Nis, Niš
  - Health Center Uzice, Užice
- United Kingdom (7):
  - Salford Royal Hospital - Northern Care Alliance NHS Foundation Trust Barnes Clinical Research Facility, Salford, Greater Manchester
  - Medicines Evaluation Unit Ltd., Wythenshawe, Greater Manchester
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich, Norfolk
  - University Hospitals Birmingham NHS Foundation Trust of Trust Headquarters Queen Elizabeth hospital Birmingham, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust Birmingham Heartlands Hospital, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Guy's and St Thomas' NHS Foundation Trust, London